CLINICAL TRIAL: NCT01139580
Title: A Multicenter, Randomized, Double-Blind Study of the Safety and Efficacy of Calcipotriene Foam, 0.005%, Versus Vehicle Foam In The Treatment Of Moderate Plaque-Type Scalp And Body Psoriasis
Brief Title: The Purpose of This Study is to Demonstrate the Safety and Effectiveness of Calcipotriene Foam in Subjects With Scalp and Body Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114743; U0267-303 (Other: Stiefel)
Record Dates: First submitted 2010-06-06; First posted 2010-06-08 (Estimated); Results first posted 2011-09-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcipotriene Foam (Experimental): Calcipotriene Foam 0.005%,
  Interventions: Drug: Calcipotriene Foam
- Vehicle Foam (Placebo Comparator): Vehicle Foam
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Calcipotriene Foam — Calcipotriene Foam 0.005%. All treatments will be administered to the skin twice daily (am-pm) for 8 weeks for subjects in this group
  Arms: Calcipotriene Foam
Drug: Vehicle Foam — Vehicle Foam. All treatments will be administered to the skin twice daily (am-pm) for 8 weeks for subjects in this group
  Arms: Vehicle Foam

SUMMARY:
The purpose of this study is to determine the safety and effectiveness in the treatment of psoriasis on the scalp and on the body.

DETAILED DESCRIPTION:
The study subjects must have moderate psoriasis of the body and scalp with an ISGA of 3 at baseline. In addition, the subjects must have an evaluable target lesion of at least 2 cm² on the body with a score of 2 or 3 for erythema, scaling and plaque. All subjects will apply Calcipotriene Foam, 0.005% or vehicle foam topically twice a day (am and pm) to all psoriatic lesions on the body and scalp. Study visits will occur at baseline (day 1) and at weeks 1, 2, 4, and 8.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures are performed.
* Male or female subjects at least 12 years old and in good general health.
* Able to complete the study and to comply with study instructions.
* Moderate plaque-type psoriasis on the body (excluding the scalp and face) defined as:

  * Plaque-type psoriasis involving 3% to 10% of total body surface area (BSA).
  * An Investigator's Static Global Assessment (ISGA) score of 3 at Baseline.
  * Identification of a target lesion (>2 cm²) on the trunk or extremities with a score of 2 or 3 (0-5 scale) for erythema, scaling and plaque thickness. Lesions on the palms/soles, knees, elbow, and intertriginous areas should not be used as the target lesion site.
* Involvement of at least 10% of the total scalp surface area with clinical signs (erythema, thickness, and scaliness) rated as moderate (3) based on the ISGA.
* Negative urine pregnancy test for females of childbearing potential. • Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are fewer than 2 years from their last menses.

Exclusion Criteria:

* Any subject who has participated in any previous calcipotriene foam clinical.
* Female who is pregnant, trying to become pregnant, or breastfeeding.
* Known allergy or other adverse reaction to calcipotriene or other vitamin D analogs; or to any component of the investigational formulations.
* History of hypercalcemia or of vitamin D toxicity.
* Other serious skin disorder or any chronic medical condition that is not well-controlled.
* Use of nonbiologic systemic anti-psoriatic therapy (eg, corticosteroids, psoralen combined with exposure to ultraviolet light A [PUVA], ultraviolet light B [UVB], retinoids, methotrexate, cyclosporine, other immunosuppressive agents) within 4 weeks prior to enrollment.
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (whichever is longer) for experimental products prior to randomization.
* Use of topical therapies that have a known beneficial effect on psoriasis, including but not limited to corticosteroids, retinoids, Vitamin D derivatives, coal tar, or anthralin, within 2 weeks prior to enrollment.
* Systemic medications for other medical conditions that are known to affect psoriasis (eg, lithium, beta adrenergic blockers) within 4 weeks prior to enrollment.
* Use of any investigational product within 4 weeks prior to enrollment, currently participating in another clinical trial, or plans to receive an investigational product during the study.
* Current drug or alcohol abuse (drug screening not required).
* Has a history of any immuno-compromizing disease.
* Any other condition that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.
* Employees of the investigator; study center; or Stiefel, a GSK company involved in the study; or an immediate family member (eg, partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (26):
  - Genova Clinical Research, Tucson, Arizona
  - Therapeutics Clinical Research Center, Inc., San Diego, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - Miami Dermatology Research Institute LLC, North Miami Beach, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Dermatology Specialists, Louisville, Kentucky
  - DermResearch, PLLC, Louisville, Kentucky
  - Henry Ford Medical Center, Detroit, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology PC, St Louis, Missouri
  - Mt. Sinai School of Medicine Div. Dermatologic & Cosmetic Surgery, New York, New York
  - Dermatology Associates of Rochester, PC, Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina
  - Group Health Associates, Cincinnatti, Ohio
  - Oregon Medical, Portland, Oregon
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Tennessee Clinical Research, Nashville, Tennessee
  - DermReserach, Inc., Austin, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Education and Research Foundation, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114743 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcipotriene Foam: Calcipotriene foam 0.005% was applied to the affected area(s) on the scalp and body twice daily (BD) for 8 weeks.
- Vehicle Foam: Vehicle foam was applied to the affected area(s) on the scalp and body BD for 8 weeks.
Period: Overall Study
Arm/Group | Calcipotriene Foam | Vehicle Foam
Started | 181 | 182
Completed | 158 | 164
Not Completed | 23 | 18
Not completed — Adverse Event | 5 | 4
Not completed — Lost to Follow-up | 9 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Used Excluded Medicine After Enrollment | 1 | 0
Not completed — Did Not Meet Exclusion Criteria | 1 | 0
Not completed — Misrandomized | 1 | 0
Not completed — Beginning Study Exclusion Treatment | 0 | 1
Not completed — Participant Randomization in Error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Calcipotriene Foam: Calcipotriene foam 0.005% was applied to the affected area(s) on the scalp and body BD for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Calcipotriene Foam | Vehicle Foam | Total
Number analyzed (Participants) | 181 | 182 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (15.3) | 44.4 (15.5) | 45.2 (15.4)
Gender [Count of Participants; unit: Participants]
  Female | 69 | 76 | 145
  Male | 112 | 106 | 218
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 3 | 9
  Black | 15 | 18 | 33
  Multiracial | 1 | 1 | 2
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0
  White | 156 | 160 | 316
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator's Static Global Assessment (ISGA) Score of Clear (0) or Almost Clear (1) for Scalp Involvement at Week 8 Using the Failure Method
Description: The investigator assessed participants with scalp psoriasis using the ISGA, scored as (as a visual average of lesions): 0, absence of disease; 1, very mild disease, lesions (L) with minimum erythema; 2, mild disease, L with light-red coloration, slight thickness, and fine, thin scale layer; 3, moderate disease, L with red coloration, moderate thickness, and a moderate scaled layer; 4, severe disease, L with red coloration, severe thickness, and a severe coarse, thick scale layer; 5, very severe disease, L with red coloration, very severe thickness, and a very severe, coarse, thick scale layer.
Time Frame: Week 8
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and dispensed study product. Missing values at Week 8 were considered to be failures. Failures were those participants who did not achieve a 2-grade improvement in IGSA score and a score of 0 or 1.
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants | 74 | 44
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With a Target Lesion Score of 0 or 1 for Erythema and at Least a 2 Grade Improvement From Baseline at Week 8
Description: Erythema is redness of the skin, caused by increased blood flow in the capillaries in the lower layers of the skin. The investigator assessed participants with erythema at target lesions using the psoriasis grading scale for target lesions (PGSTL). PGSTL scores: 0, no evidence of erythema, hyperpigmentation may be present; 1, faint erythema; 2, light-red coloration; 3, moderate red coloration; 4, bright-red coloration; 5, dusky to deep red coloration.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants | 42 | 30

3. Secondary Outcome: Number of Participants With a Target Lesion Score of 0 or 1 for Scaling and at Least a 2 Grade Improvement From Baseline at Week 8
Description: Scaling of the skin is the loss of the outer layer of the epidermis in scale-like flakes. The investigator assessed participants with scaling at target lesions using the psoriasis grading scale for target lesions (PGSTL). PGSTL scores: 0, no evidence of scaling; 1, minimal, occasional fine scale over less than 5% of the lesion; 2, mild, fine scales predominate; 3, moderate, coarse scales predominate; 4 marked, thick non-tenacious scale predominates; 5 severe, very thick tenacious scale predominates.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants | 53 | 38

4. Primary Outcome: Number of Participants With an ISGA Score of Clear (0) or Almost Clear (1) for Scalp Involvement at Week 8 Using Last Observation Carried Forward (LOCF)
Description: as for outcome 1
Time Frame: Week 8
Population: ITT Population. Missing values were imputed using LOCF (i.e., the last available observation, including Baseline, for a participant will be used to estimate subsequent missing data points).
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants | 75 | 45
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants With a Target Lesion Score of 0 or 1 for Plaque Thickness at Week 8
Description: Psoriasis is a noncontagious skin disorder, most often appearing as inflamed, thickened skin covered with silvery white scales on the scalp, trunk, and limbs. The investigator assessed participants with plaque thickness at target lesions using the PGSTL scores: 0, no elevation over normal skin; 1, possible but difficult to ascertain whether there is a slight elevation above normal skin; 2, slight but definite elevation, edges are indistinct or sloped; 3, moderate elevation with rough or sloped edges; 4, marked elevation with hard or sharp edges; 5, very marked elevation with hard sharp edges.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants | 67 | 53

6. Secondary Outcome: Number of Participants With an ISGA Score of Clear (0) or Almost Clear (1) for Body Involvement at Week 8
Description: The investigator assessed participants with psoriasis with body involvement using the ISGA, scored as: 0, clear, minor residual discoloration, no erythema, scaling, or plaque thickness; 1, almost clear, occasional fine scale, faint erythema, and barely perceptible plaque thickness; 2, mild, fine scales predominate with light-red coloration and mild plaque thickness; 3, moderate, coarse scales predominate with moderate red coloration and plaque thickness; 4 severe, thick tenacious scale predominates with deep red coloration and severe plaque thickness. Scores are a visual average of lesions.
Time Frame: Week 8
Population: ITT Population. Data were analyzed using the failure and LOCF methods.
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 181 | 182
participants
  Failure method | 32 | 28
  LOCF | 33 | 28

ADVERSE EVENTS:
Arm/Group | Calcipotriene Foam | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 1/181 | 3/182
Other Adverse Events (participants affected / at risk) | 25/181 | 17/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriene Foam (N=181) | Vehicle Foam (N=182)
Chest discomfort (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriene Foam (N=181) | Vehicle Foam (N=182)
Application site pruritus (General disorders) | 7 | 7
Application site pain (General disorders) | 8 | 5
Application site erythema (General disorders) | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Nasopharyngitis (Infections and infestations) | 0 | 5
Application site dermatitis (General disorders) | 4 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.